CLINICAL TRIAL: NCT02005783
Title: Adjuvant Treatment of EC/TC Versus EC/TC Plus Danggui Buxue Decoction in Breast Cancer：A Prospective, Randomized Trial
Brief Title: Study of Danggui Buxue Decoction in Preventing Neutropenia
Acronym: DIPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Kunwei Shen, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RJBC1302
Record Dates: First submitted 2013-12-04; First posted 2013-12-09 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-05

CONDITIONS: Grade 3/4 Neutropenia; Febrile Neutropenia
Keywords: incidence of grade 3/4 neutropenia; incidence of febrile neutropenia; time to neutropenia recovery; safety
MeSH Terms: conditions — Febrile Neutropenia | interventions — danggui buxue decoction; Epirubicin; Cyclophosphamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DBD arm (Experimental): Epirubicin: 90mg/m2, d1, q3w*4 Cyclophosphamide: 600mg/m2, d1, q3w*4 DBD: one dose of medicine twice per day, orally OR; Docetaxel: 75mg/m2, d1, q3w*4 Cyclophosphamide: 600mg/m2, d1, q3w*4 DBD: one dose of medicine twice per day, orally
  Interventions: Drug: DBD; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Docetaxel
- EC/TC (Other): Epirubicin: 90mg/m2, d1, q3w*4 Cyclophosphamide: 600mg/m2, d1, q3w*4 OR; Docetaxel: 75mg/m2, d1, q3w*4 Cyclophosphamide: 600mg/m2, d1, q3w*4
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Docetaxel

INTERVENTIONS:
Drug: DBD — DBD:one dose of medicine twice per day, orally
  Other Names: Danggui Buxue Decoction
  Arms: DBD arm
Drug: Epirubicin — Epirubicin:90mg/m2, d1, q3w*4
Drug: Cyclophosphamide — Cyclophosphamide:600mg/m2, d1, q3w*4
Drug: Docetaxel — Docetaxel:75mg/m2, d1, q3w*4

SUMMARY:
To evaluate EC/TC (epirubicin and cyclophosphomide or docetaxel and cyclophosphomide) with EC/TC plus DBD (Danggui Buxue Decoction) in adjuvant treatment of breast cancer patients. The aim is to evaluate whether DBD can decrease the incidence of grade 3/4 neutropenia induced by EC/TC regimen during chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Women aged ≥18 years and < 70 years; Histologically confirmed invasive breast cancer by core needle biopsy, suggested to receive EC/TC regiments for adjuvant chemotherapy by MDT; Leukocyte ≥ 3*109/L; Neutrophil ≥ 1.5*109/L; PLT ≥ 100*109/L; Serum AST/SGOT or ALT/AGPT ≤ 2.5 times of upper limit of normal (UNL) range Serum creatinine/BUN ≤ upper limit of normal (UNL) range; No dysphagia, be able to take the Danggui Buxue Decoction(DBD) Written informed consent according to the local ethics committee requirements. Has ECOG Performance Score 0-1;

Exclusion Criteria:

Metastatic breast cancer; Family history of endometrial cancer or any other kind of gynecologic cancer; Patients with severe co-morbidity that indicate intolerant to adjuvant chemotherapy; patients with psychiatric disorder or other diseases leading to incompliance to the therapy; Known severe hypersensitivity to any drugs in this study; Prior adjuvant chemotherapy of any kind cancer; Hematologic disorders relative to aplasia

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
incidence of grade 3/4 neutropenia | 3 weeks
  To compare the incidence of grade 3/4 neutropenia between EC/TC arm and EC/TC plus DBD arm in breast cancer adjuvant chemotherapy.

SECONDARY OUTCOMES:
times of grade 3/4 neutropenia per cycle of chemotherapy | 3 weeks
  To compare the times of grade 3/4 neutropenia per cycle of chemotherapy between EC/TC arm and EC/TC plus DBD arm in breast cancer adjuvant chemotherapy.
incidence of febrile neutropenia | 3 weeks
  to compare incidence of febrile neutropenia between EC/TC arm and EC/TC plus DBD arm in breast cancer adjuvant chemotherapy.
the time to neutropenia recovery | 2 months
  to compare the time to neutropenia recovery between EC/TC arm and EC/TC plus DBD arm in breast cancer adjuvant chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Kunwei Shen, Dr, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China